CLINICAL TRIAL: NCT01944774
Title: A Multi-Center, Randomized, Double-Blind, Parallel Comparative, Phase II Study to Evaluate the Efficacy and Safety of Intravenous Infusion With Nemonoxacin Versus Moxifloxacin in Treating Adult Patients With Community-Acquired Pneumonia
Brief Title: Study to Evaluate the Efficacy and Safety of Intravenous Infusion With Nemonoxacin Malate Sodium Chloride
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Collaborators: QPS-Qualitix (Industry); R&G Pharma Studies Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-873870-C-5
Record Dates: First submitted 2013-08-26; First posted 2013-09-18 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2015-02

CONDITIONS: Pneumonia
Keywords: Moxifloxacin
MeSH Terms: conditions — Pneumonia | interventions — nemonoxacin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nemonoxacin 500 mg (Experimental): Nemonoxacin 500mg/250mL.
  Interventions: Drug: Nemonoxacin 500 mg
- Nemonoxacin 650 mg (Experimental): Nemonoxacin 650 mg/325mL
  Interventions: Drug: Nemonoxacin 650 mg
- Moxifloxacin 400 mg (Active Comparator): Moxifloxacin 400mg/250mL
  Interventions: Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: Nemonoxacin 500 mg — IV Infusion, once daily for 7~14 days
  Other Names: Taigexyn infusion solution
  Arms: Nemonoxacin 500 mg
Drug: Nemonoxacin 650 mg — IV Infusion, once daily for 7~14 days
  Other Names: Taigexyn infusion solution
  Arms: Nemonoxacin 650 mg
Drug: Moxifloxacin 400 mg — IV Infusion, once daily for 7~14 days
  Other Names: Moxifloxacin infusion solution
  Arms: Moxifloxacin 400 mg

SUMMARY:
The purpose of this study is to Evaluate the Efficacy, safety and pharmacokinetics of Intravenous Nemonoxacin Compared with Intravenous Moxifloxacin in Adult Patients with community-acquired pneumonia (CAP).

DETAILED DESCRIPTION:
Community-acquired Pneumonia (CAP) remains a leading cause of death in both developing and developed countries. In the choice of antibacterial agents used to treat CAP, fluoroquinolones have received considerable attention because of their wide spectrum of bactericidal activity. TG-873870 (Nemonoxacin), a non-fluorinated quinolone (NFQ), is a selective bacterial topoisomerase inhibitor.

This study will Evaluate the clinical efficacy, microbiological efficacy and safety of Intravenous Nemonoxacin compared with Intravenous Moxifloxacin in adult patients with community-acquired pneumonia.

Besides, the pharmacokinetics (PK) of Nemonoxacin in adult patients with CAP after continuous IV Infusion and the pharmacokinetic (PK)/pharmacodynamic (PD)are to be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18 and 75;
2. Weighs between 40 ~ 100 kg, and BMI ≥ 18 kg/m2;
3. Must have a clinical diagnosis of CAP
4. Chest X-ray and /or CT scan show new or persist/progressive infiltrates
5. Patients with PORT/PSI score II, III or IV.
6. If female, non-lactating and at no risk or pregnancy (post-menopausal or must use adequate birth control)
7. The patient is able to receive an intravenous infusion of the drug .

Exclusion Criteria:

1. Patients with PORT/PSI score I or VI.
2. Severe CAP is present if a patient needs invasive mechanical ventilation or requires vasopressors.
3. Known or suspected severe bronchiectasis, cystic fibrosis, active pulmonary tuberculosis or infection with other mycobacteria or fungi, known bronchial obstruction, a history of post-obstructive pneumonia, other confounding respiratory diseases, such as lung cancer, malignancy metastatic to the lungs, lung abscess, empyema, suspected aspiration pneumonia due to vomiting, or non-bacterial respiratory infection (chronic obstructive pulmonary disease [COPD] is not exclusionary)
4. Clinically significant conduction or other abnormality on 12-lead ECG, or QTc interval
5. Potassium is < 3.5 mmol/L
6. Any known disease that seriously affect the immune system
7. Active hepatitis or decompensated cirrhosis;
8. Have used quinolones or fluoroquinolones within 14 days before enrollment
9. Patients who are being or will be on a long-term medication of steroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LiWen Chang, Study Director — Taigenbiotech
Locations (2):
- Institute of Antibiotics, Huashan Hospital, Fundan University, Shanghai, China
- Far eastern memorial hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wu XJ, Zhang J, Guo BN, Zhang YY, Yu JC, Cao GY, Chen YC, Zhu DM, Ye XY, Wu JF, Shi YG, Chang LW, Chang YT, Tsai CY. Pharmacokinetics and pharmacodynamics of multiple-dose intravenous nemonoxacin in healthy Chinese volunteers. Antimicrob Agents Chemother. 2015 Mar;59(3):1446-54. doi: 10.1128/AAC.04039-14. Epub 2014 Dec 22. PMID 25534726
- [Derived] Cao GY, Zhang J, Zhang YY, Guo BN, Yu JC, Wu XJ, Chen YC, Wu JF, Shi YG. Safety, tolerability, and pharmacokinetics of intravenous nemonoxacin in healthy chinese volunteers. Antimicrob Agents Chemother. 2014 Oct;58(10):6116-21. doi: 10.1128/AAC.02972-14. Epub 2014 Aug 4. PMID 25092690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 41 research centers in China and Taiwan. Among these, 11 research centers did not enroll participants. 207 subjects were randomly enrolled in the 30 research centers.
Period: Overall Study
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Started | 69 | 68 | 70
Received Treatment | 68 | 67 | 70
Completed | 63 | 60 | 62
Not Completed | 6 | 8 | 8
Not completed — Withdrawal by Subject | 2 | 3 | 3
Not completed — Adverse Event | 3 | 2 | 3
Not completed — Lack of Efficacy | 1 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: mITT population: Subjects who were screened and randomized, received at least one complete dose of the drug (Nemonoxacin or Moxifloxacin), met the minimal disease criteria (inclusion criteria 4, 5 and 7), and was evaluated at least once for clinical efficacy .
Groups:
- Total: Total of all reporting groups
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg | Total
Number analyzed (Participants) | 67 | 64 | 64 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (15.33) | 53.5 (14.21) | 51.5 (16.00) | 52.6 (15.14)
Age, Customized [Number; unit: participants]
  ≧18 and <30 years | 6 | 4 | 10 | 20
  ≧30 and < 40 years | 9 | 8 | 9 | 26
  ≧40 and < 50 years | 10 | 12 | 8 | 30
  ≧50 and < 60 years | 16 | 15 | 11 | 42
  ≧60 and < 70 years | 16 | 17 | 17 | 50
  ≧70 and < 76 years | 10 | 8 | 9 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 23 | 71
  Male | 42 | 41 | 41 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 67 | 64 | 64 | 195
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Nationality [Number; unit: participants]
  Han | 62 | 61 | 61 | 184
  Minority ethnic groups | 3 | 2 | 1 | 6
  Taiwan Aborigines | 0 | 0 | 1 | 1
  Unknown | 2 | 1 | 1 | 4
Height [Mean (Standard Deviation); unit: cm] | 163.5 (7.08) | 164.2 (8.65) | 164.7 (8.68) | 164.1 (8.13)
Weight [Mean (Standard Deviation); unit: kg] | 60.0 (8.45) | 63.5 (12.94) | 64.3 (11.81) | 62.5 (11.29)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.5 (3.01) | 23.4 (3.44) | 23.6 (3.29) | 23.1 (3.27)
PORT/PSI score [Number; unit: participants] — The pneumonia severity index PSI or PORT Score is a clinical prediction rule that medical practitioners use to calculate the probability of morbidity and mortality among patients with CAP. Point values are given for various parameters of demographics, comorbidity, physical exam fndings, lab and radiographic findings. The total PSI score places a given patient into one of 5 risk classes. Classes I, II, and III are at low risk for death, and may be considered for outpatient treatment. Risk classes IV and V should be hospitalized and even an intensive care should be considered.
  participants
    Class II | 31 | 33 | 30 | 94
    Class III | 34 | 28 | 29 | 91
    Class IV | 2 | 3 | 5 | 10
Smoking status [Number; unit: participants]
  Never smoked | 45 | 32 | 43 | 120
  Former smoker (abstinent for a minimum of 2 years) | 8 | 8 | 4 | 20
  Current smoker or smoked within the past 2 years | 14 | 24 | 17 | 55
Drinking status [Number; unit: participants]
  Lifetime abstainer | 54 | 41 | 39 | 134
  Former drinker | 4 | 3 | 7 | 14
  Current drinker | 9 | 20 | 18 | 47

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Clinical Cure Rate of Two Doses of Intravenously Infused Nemonoxacin Malate Sodium Chloride Injection at Visit 4 in the mITT Population
Description: The primary efficacy endpoint of this study was to evaluate whether the clinical cure rate of Nemonoxacin malate sodium chloride is non-inferior to that of Moxifloxacin at visit 4 in the mITT population. At visit 4, the Investigator would assess changes in the symptoms/signs/laboratory tests and chest X-rays/or CT scans associated with this infection, and determined the clinical efficacy in the subjects. The clinical efficacy of the study group and the control group was calculated according to the proportion and percentage of overall clinically cured and clinically ineffective patients in the treatment groups. If the lower limit of the 90% confidence interval for the difference in the clinical cure rate between the study drug and the control drug was larger than -15%, it would be established that the efficacy of Nemonoxacin malate sodium chloride injection was not inferior to that of Moxifloxacin Hydrochloride Sodium Chloride Injection in the treatment of moderate to severe adult CAP.
Time Frame: Visit 1 (baseline, day -1~1) to Visit 4 (7-14 days after stopping the drug)
Population: Subjects in the ITT population that met the minimal disease criteria, and was evaluated for clinical efficacy at least once were enrolled into the mITT population.
Measure: Number; unit: participants
Groups:
- Nemonoxacin 500 mg: Nemonoxacin 500mg/250mL. Nemonoxacin 500 mg: IV Infusion, once daily for 7~14 days
- Nemonoxacin 650 mg: Nemonoxacin 650 mg/325mL Nemonoxacin 650 mg: IV Infusion, once daily for 7~14 days
- Moxifloxacin 400 mg: Moxifloxacin 400mg/250mL Moxifloxacin 400 mg: IV Infusion, once daily for 7~14 days
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 67 | 64 | 64
participants
  Success | 60 | 58 | 59
  Fail | 7 | 4 | 2
  Not evaluable | 0 | 2 | 3
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Non-Inferiority or Equivalence — Clinical success rate was assumed for the experimental group (Nemonoxacin 500mg) and the control group (Moxifloxacin 400mg) were both 88%. The non-inferiority margin was defined as 15%, one-sided significance value was 0.05 (one-tailed α=0.05), power was 80%, and the assignment ratio was 1:1:1; p = 0.133, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.291, 95% CI 2-sided [0.058 to 1.457]
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Non-Inferiority or Equivalence — Clinical success rate was assumed for the experimental group (Nemonoxacin 650mg) and the control group (Moxifloxacin 400mg) were both 88%. The non-inferiority margin was defined as 15%, one-sided significance value was 0.05 (one-tailed α=0.05), power was 80%, and the assignment ratio was 1:1:1; p = 0.423, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.492, 95% CI 2-sided [0.087 to 2.788]

2. Secondary Outcome: Difference in the Clinical Cure Rate of Two Doses of Intravenously Infused Nemonoxacin Malate Sodium Chloride Injection at Visit 4 in the Clinically Evaluable (CE) Population
Description: The primary efficacy endpoint of this study was to evaluate whether the clinical cure rate of Nemonoxacin malate sodium chloride is non-inferior to that of Moxifloxacin at visit 4 in the CE population. At visit 4, the Investigator would assess changes in the symptoms/signs/laboratory tests and chest X-rays/or CT scans associated with this infection, and determined the clinical efficacy in the subjects. The clinical efficacy of the study group and the control group was calculated according to the proportion and percentage of overall clinically cured and clinically ineffective patients in the treatment groups. If the lower limit of the 90% confidence interval for the difference in the clinical cure rate between the study drug and the control drug was larger than -15%, it would be established that the efficacy of Nemonoxacin malate sodium chloride injection was not inferior to that of Moxifloxacin Hydrochloride Sodium Chloride Injection in the treatment of moderate to severe adult CAP.
Time Frame: Visit 1 (baseline, day -1~1) to Visit 4 (7-14 days after stopping the drug)
Population: Subjects in the mITT population that conformed to the protocol analysis plan with no major violation to the protocol were enrolled into the CE population.
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 63 | 59 | 60
participants
  Success | 56 | 56 | 58
  Not evaluable | 7 | 3 | 2
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.118, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.276, 95% CI 2-sided [0.055 to 1.385]
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.636, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.644, 95% CI 2-sided [0.104 to 3.999]

3. Secondary Outcome: Difference in the Clinical Cure Rate of Two Doses of Intravenously Infused Nemonoxacin Malate Sodium Chloride Injection at Visit 3 in the mITT Population
Description: The primary efficacy endpoint of this study was to evaluate whether the clinical cure rate of Nemonoxacin malate sodium chloride is non-inferior to that of Moxifloxacin at visit 3 in the mITT population. At visit 3, the Investigator would assess changes in the symptoms/signs/laboratory tests and chest X-rays/or CT scans associated with this infection, and determined the clinical efficacy in the subjects. The clinical efficacy of the study group and the control group was calculated according to the proportion and percentage of overall clinically cured and clinically ineffective patients in the treatment groups. If the lower limit of the 90% confidence interval for the difference in the clinical cure rate between the study drug and the control drug was larger than -15%, it would be established that the efficacy of Nemonoxacin malate sodium chloride injection was not inferior to that of Moxifloxacin Hydrochloride Sodium Chloride Injection in the treatment of moderate to severe adult CAP.
Time Frame: Visit 1 (baseline, day -1~1) to Visit 3 (Within 24 hours after stopping the drug)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 67 | 64 | 64
participants
  Success | 61 | 60 | 59
  Fail | 4 | 4 | 2
  Not evaluable | 2 | 0 | 3
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.456, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.517, 95% CI 2-sided [0.091 to 2.930]
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.445, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.508, 95% CI 2-sided [0.090 to 2.883]

4. Secondary Outcome: Difference in the Clinical Cure Rate of Two Doses of Intravenously Infused Nemonoxacin Malate Sodium Chloride Injection at Visit 3 in the CE Population
Description: The primary efficacy endpoint of this study was to evaluate whether the clinical cure rate of Nemonoxacin malate sodium chloride is non-inferior to that of Moxifloxacin at visit 3 in the CE population. At visit 3, the Investigator would assess changes in the symptoms/signs/laboratory tests and chest X-rays/or CT scans associated with this infection, and determined the clinical efficacy in the subjects. The clinical efficacy of the study group and the control group was calculated according to the proportion and percentage of overall clinically cured and clinically ineffective patients in the treatment groups. If the lower limit of the 90% confidence interval for the difference in the clinical cure rate between the study drug and the control drug was larger than -15%, it would be established that the efficacy of Nemonoxacin malate sodium chloride injection was not inferior to that of Moxifloxacin Hydrochloride Sodium Chloride Injection in the treatment of moderate to severe adult CAP.
Time Frame: Visit 1 (baseline, day -1~1) to Visit 3 (Within 24 hours after stopping the drug)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 63 | 59 | 60
participants
  Success | 58 | 56 | 56
  Fail | 4 | 3 | 2
  Not evaluable | 1 | 0 | 2
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.458, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.518, 95% CI 2-sided [0.091 to 2.941]
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.664, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.667, 95% CI 2-sided [0.107 to 4.144]

5. Secondary Outcome: Subject Number for Microbiologically Cured and Failure at Visit 4 in b-mITT (Bacteriological mITT) Population
Description: Microbiological efficacy at visits 4 would be determined by assessing the identification results from the central laboratory. Subjects must satisfy at least one of the following in order to be evaluated for the microbiological efficacy:
  1. Subjects whose respiratory culture from visit 1 was positive;
  2. Subjects whose blood culture from visit 1 was positive.
  The microbiological efficacy at Visit 4 and treatment group (determined by each subject) was determined by the number and percentage of microbiological success subjects. The difference in bacteriological success between Nemonoxacin malate sodium chloride injection and Moxifloxacin Hydrochloride Sodium Chloride Injection was tested using the logistic regression model.
Time Frame: Visit 1 (baseline, day -1~1) to Visit 4 (7-14 days after stopping the drug)
Population: Subjects in the mITT population whose bacterial culture yielded at least one baseline bacterial isolate were enrolled into the b-mITT population.
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 24 | 19 | 17
participants
  Success | 21 | 17 | 16
  Failure | 3 | 1 | 0
  Not evaluable | 0 | 1 | 1
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.959, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.000 — The 2-sided 95% confidence interval of OR is (<0.001, >999.999)
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.961, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.000 — The 2-sided 95% confidence interval of OR is (<0.001, >999.999)

6. Secondary Outcome: Subject Number for Microbiologically Cured and Failure at Visit 4 in BE (Bacteriological Evaluable) Population
Description: as for outcome 5
Time Frame: Visit 1 (baseline, day -1~1) to Visit 4 (7-14 days after stopping the drug)
Population: Subjects in the b-mITT population who conformed to the protocol analysis plan with no major violation to the protocol were enrolled into the BE population.
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 23 | 19 | 16
participants
  Success | 20 | 17 | 15
  Failure | 3 | 1 | 0
  Not evaluable | 0 | 1 | 1
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.960, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.000 — The 2-sided 95% confidence interval of OR is (<0.001, >999.999)
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.962, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.000 — The 2-sided 95% confidence interval of OR is (<0.001, >999.999)

7. Secondary Outcome: Subject Number for Microbiologically Cured and Failure at Visit 3 in b-mITT (Bacteriological mITT) Population
Description: Microbiological efficacy at visits 3 would be determined by assessing the identification results from the central laboratory. Subjects must satisfy at least one of the following in order to be evaluated for the microbiological efficacy:
  1. Subjects whose respiratory culture from visit 1 was positive;
  2. Subjects whose blood culture from visit 1 was positive.
  The microbiological efficacy at Visit 3 and treatment group (determined by each subject) was determined by the number and percentage of microbiological success subjects. The difference in bacteriological success between Nemonoxacin malate sodium chloride injection and Moxifloxacin Hydrochloride Sodium Chloride Injection was tested using the logistic regression model.
Time Frame: Visit 1 (baseline, day -1~1) to Visit 3 (Within 24 hours after stopping the drug)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 24 | 19 | 17
participants
  Success | 22 | 18 | 16
  Failure | 2 | 1 | 0
  Not evaluable | 0 | 0 | 1
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.950, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.000 — The 2-sided 95% confidence interval of OR is (<0.001, >999.999)
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.962, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.000 — The 2-sided 95% confidence interval of OR is (<0.001, >999.999)

8. Secondary Outcome: Subject Number for Microbiologically Cured and Failure at Visit 3 in BE (Bacteriological Evaluable) Population
Description: as for outcome 7
Time Frame: Visit 1 (baseline, day -1~1) to Visit 3 (Within 24 hours after stopping the drug)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 23 | 19 | 16
participants
  Success | 21 | 18 | 16
  Failure | 2 | 1 | 0
  Not evaluable | 0 | 0 | 0
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.949, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.000 — The 2-sided 95% confidence interval of OR is (<0.001, >999.999)
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.962, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.000 — The 2-sided 95% confidence interval of OR is (<0.001, >999.999)

9. Secondary Outcome: Subject Number of Success and Failure in Overall Efficacy at Visit 4 in b-mITT (Bacteriological mITT) Population
Description: Only subjects whose bacterial culture from visit 1 was positive would be evaluated for the overall efficacy. The overall efficacy (cured or ineffective) at Visit 4 and treatment group (determined by each subject) was determined by the number and percentage of subjects. The difference in bacteriological success between Nemonoxacin malate sodium chloride injection and Moxifloxacin Hydrochloride Sodium Chloride Injection was tested using the logistic regression model.
Time Frame: Visit 1 (baseline, day -1~1) to Visit 4 (7-14 days after stopping the drug)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 24 | 19 | 17
participants
  Success | 21 | 17 | 16
  Failure | 3 | 2 | 1
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.491, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.438, 95% CI 2-sided [0.042 to 4.609]
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.619, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.531, 95% CI 2-sided [0.044 to 6.444]

10. Secondary Outcome: Subject Number of Success and Failure in Overall Efficacy at Visit 4 in BE (Bacteriological Evaluable) Population
Description: as for outcome 9
Time Frame: Visit 1 (baseline, day -1~1) to Visit 4 (7-14 days after stopping the drug)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 23 | 19 | 16
participants
  Success | 20 | 17 | 15
  Failure | 3 | 2 | 1
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.501, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.444, 95% CI 2-sided [0.042 to 4.708]
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.656, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.567, 95% CI 2-sided [0.047 to 6.895]

11. Secondary Outcome: Subject Number of Success and Failure in Overall Efficacy at Visit 3 in b-mITT (Bacteriological mITT) Population
Description: Only subjects whose bacterial culture from visit 1 was positive would be evaluated for the overall efficacy. The overall efficacy (cured or ineffective) at Visit 3 and treatment group (determined by each subject) was determined by the number and percentage of subjects. The difference in bacteriological success between Nemonoxacin malate sodium chloride injection and Moxifloxacin Hydrochloride Sodium Chloride Injection was tested using the logistic regression model.
Time Frame: Visit 1 (baseline, day -1~1) to Visit 3 (Within 24 hours after stopping the drug)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 24 | 19 | 17
participants
  Success | 22 | 17 | 15
  Failure | 2 | 2 | 1
  Unevaluable | 0 | 0 | 1
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.807, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.733, 95% CI 2-sided [0.061 to 8.832]
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.656, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.567, 95% CI 2-sided [0.047 to 6.895]

12. Secondary Outcome: Subject Number of Success and Failure in Overall Efficacy at Visit 3 in BE (Bacteriological Evaluable) Population
Description: as for outcome 11
Time Frame: Visit 1 (baseline, day -1~1) to Visit 3 (Within 24 hours after stopping the drug)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 23 | 19 | 16
participants
  Success | 21 | 17 | 15
  Failure | 2 | 2 | 1
Statistical Analysis 1: Comparison: Nemonoxacin 500 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.779, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.700, 95% CI 2-sided [0.058 to 8.445]
Statistical Analysis 2: Comparison: Nemonoxacin 650 mg vs Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.656, Regression, Logistic — Only P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.567, 95% CI 2-sided [0.047 to 6.895]

ADVERSE EVENTS:
Time Frame: The whole study period: from Screening Vsit (day -1~1) to Visit 4 (7-14 days after stopping the drug)
Arm/Group | Nemonoxacin 500 mg | Nemonoxacin 650 mg | Moxifloxacin 400 mg
Serious Adverse Events (participants affected / at risk) | 3/68 | 1/67 | 1/70
Other Adverse Events (participants affected / at risk) | 51/68 | 41/67 | 33/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemonoxacin 500 mg (N=68) | Nemonoxacin 650 mg (N=67) | Moxifloxacin 400 mg (N=70)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Possibly related to the study drug
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Possibly related to the study drug
Worsening of congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Possibly unrelated to the study drug
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) — Possibly unrelated to the study drug for SAE occurred in subjects in the Nemonoxacin 650mg study group and definitely unrelated to the study drug for for SAE occurred in subjects in the Nemonoxacin 500mg study group
Lung neoplasm malignant (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Definitely unrelated to the study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemonoxacin 500 mg (N=68) | Nemonoxacin 650 mg (N=67) | Moxifloxacin 400 mg (N=70)
Alanine aminotransferase increased (Investigations) | 4 (4) | 14 (14) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 11 (11) | 4 (4)
White blood cell count decreased (Investigations) | 3 (3) | 5 (6) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 5 (5) | 2 (2)
Red blood cells urine positive (Investigations) | 2 (2) | 3 (3) | 2 (2)
Red blood cell count decreased (Investigations) | 2 (2) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (3) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 3 (3) | 2 (3)
Blood albumin decreased (Investigations) | 3 (4) | 1 (1) | 2 (2)
Blood potassium decreased (Investigations) | 2 (2) | 3 (3) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 2 (2) | 1 (1)
Haematocrit decreased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Neutrophil percentage decreased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 2 (2) | 2 (2)
White blood cell count increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Platelet count increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Protein total decreased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Monocyte percentage increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Monocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte percentage increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Mean cell haemoglobin concentration decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Mean cell haemoglobin concentration increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prealbumin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eosinophil percentage increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil percentage increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram ST-T change (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave amplitude decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Total bile acids increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 11 (20) | 11 (25) | 4 (5)
Infusion site pruritus (General disorders) | 8 (23) | 8 (25) | 3 (8)
Infusion site pain (General disorders) | 4 (11) | 3 (8) | 2 (10)
Infusion site discomfort (General disorders) | 4 (16) | 1 (1) | 0 (0)
Infusion site rash (General disorders) | 2 (2) | 2 (2) | 0 (0)
Infusion site swelling (General disorders) | 2 (5) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Flushing (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Supraventricular arrhythmias (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Cardiac conduction disorders (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Palpitation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Chest discomfort (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea manuum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Gait disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Altered visual depth perception (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (4) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Rheumatoid arthritis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0)
Renal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenias NEC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI needs to inform sponsor and asks for permission before he/she discusses or publishes trial results after the trial is completed.